CLINICAL TRIAL: NCT02491125
Title: Effect of Prebiotic Fibre on Intestinal Health and Functioning
Brief Title: The Effect of Prebiotics on Gastrointestinal Functioning and Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NL52300.068.15
Record Dates: First submitted 2015-03-23; First posted 2015-07-07 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2018-10

CONDITIONS: Change of Transit or Circulation; Obesity
MeSH Terms: conditions — Obesity | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 12 weeks placebo maltodextrin 15g/day ( 5 g in beverage, to be consumed three times a day)
  Interventions: Dietary Supplement: Placebo
- soluble wheat bran fibre (Experimental): 12 weeks soluble wheat bran fibre 15g/day (5 g in beverage, to be consumed three times a day)
  Interventions: Dietary Supplement: soluble wheat bran fibre

INTERVENTIONS:
Dietary Supplement: soluble wheat bran fibre — 12 weeks daily intake of 15g of soluble wheat bran fibre
  Arms: soluble wheat bran fibre
Dietary Supplement: Placebo — 12 weeks daily intake of 15g of maltodextrin
  Other Names: Maltodextrin
  Arms: Placebo

SUMMARY:
The study will investigate the effect of cereal based prebiotic fibres on intestinal health and functioning and host metabolism.

DETAILED DESCRIPTION:
A human dietary intervention study will be performed in overweight to obese subjects with a slow gastrointestinal transit time comparing the effects of a soluble prebiotic fibre vs. placebo on gut health, including gut microbiota composition, gastrointestinal transit time, metabolic health and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Overweight to obese men and women (BMI ≥ 25 kg/m2 <35 kg/m2)
* Aged 20-50 years
* Caucasian
* Normal fasting glucose (<6.1 mmol/L.)
* Normal blood pressure (systolic blood pressure 100-140 mmHg, diastolic blood pressure 60-90 mmHg)
* Weight stable in last 3 months (±2 kg)
* A low defecation frequency, <4 times/week and no constipation or underlying pathology, as determined by gastro-intestinal questionnaires).
* A slow whole gut transit (>35h)

Exclusion Criteria:

* Woman lactating, pregnant (where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test) or (post)-menopausal
* Regular smokers
* People with intensive fitness training, eg. athletes (≥3 per week ≥ 1 hour training)
* Diabetes Mellitus (defined as FPG ≥ 7.0 mmol/l and or 2h PG ≥ 11.1 mmol/l)
* Gastro-intestinal diseases or abdominal surgery, cardiovascular diseases, cancer, liver or kidney malfunctioning (determined based on ALAT and creatinine levels, respectively) disease with a life expectation shorter than 5 years
* Following a hypocaloric diet
* Gluten intolerance
* Regular use of laxation products, or use of antibiotics, probiotics or prebiotics 3 months prior to the start of the study
* More than 2 symptoms occurring over a period of 12 weeks in the preceding 12 months such as

  1. Straining in >1/4 defecations;
  2. Lumpy or hard stools in >1/4 defecations;
  3. Sensation of incomplete evacuation in >1/4 defecations;
  4. Sensation of anorectal obstruction/blockade in >1/4 defecations
  5. Manual maneuvers to facilitate >1/4 defecations (e.g., digital evacuation, support of the pelvic floor); and/or
  6. <3 defecations/week
* Current use of medication interfering with study intervention or interfering with study endpoints/hypotheses
* Not to be able to understand the study information
* Blood donation 2 months prior to the study and during the study
* Participation in other studies

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Whole gut transit time [hours] | measured at baseline at week 1 and directly after the 12 week supplementation
  Whole gut transit time as measured by radio-opaque marker method

SECONDARY OUTCOMES:
Gastric emptying [min] | measured at baseline at week 1 and directly after the 12 week supplementation
  Gastric emptying measured by isotope breath test
Oro-cecal transit time [min] | measured at baseline at week 1 and directly after the 12 week supplementation
  Oro-cecal transit time measured by hydrogen breath test
Defecation frequency (bowel movement per day) | measured at baseline at week 1 and directly after the 12 week supplementation
  Defecation frequency as measured via questionnaire
Energy expenditure | measured at baseline at week 1 and directly after the 12 week supplementation
  Energy expenditure measured by indirect calorimetry
Substrate oxidation | measured at baseline at week 1 and directly after the 12 week supplementation
  Fat and carbohydrate oxidation measured by indirect calorimetry
Plasma inflammatory cytokines Interleukin-6,8 and 1 (pg/ml) | measured at baseline at week 1 and directly after the 12 week supplementation
  IL-6, IL8,IL-1 measured by enzyme linked immunosorbent assay
Adipose tissue gene expression | measured at baseline at week 1 and directly after the 12 week supplementation
  Adipose tissue gene expression measured by quantitative real time polymerase chain reaction
Gut permeability | measured at baseline at week 1 and directly after the 12 week supplementation
  Gut permeability as measured by multi sugar assay
Microbiota composition | measured at baseline at week 1 and directly after the 12 week supplementation
  Microbiota composition as measured by illumina sequencing in feces
Fecal Short chain fatty acid concentrations | measured at baseline at week 1 and directly after the 12 week supplementation
  Fecal Short chain fatty acid concentrations measured by ion exchange chromatography with conductivity detection
Plasma short chain fatty acid concentrations | measured at baseline at week 1 and directly after the 12 week supplementation
  Plasma short chain fatty acid concentrations measured by liquid chromatography-mass spectrometry

REFERENCES:
- [Derived] Muller M, Hermes GDA, Emanuel E C, Holst JJ, Zoetendal EG, Smidt H, Troost F, Schaap FG, Damink SO, Jocken JWE, Lenaerts K, Masclee AAM, Blaak EE. Effect of wheat bran derived prebiotic supplementation on gastrointestinal transit, gut microbiota, and metabolic health: a randomized controlled trial in healthy adults with a slow gut transit. Gut Microbes. 2020 Nov 9;12(1):1704141. doi: 10.1080/19490976.2019.1704141. Epub 2020 Jan 25. PMID 31983281